CLINICAL TRIAL: NCT06985511
Title: Assessment of Marginal Bone Loss and Anterior Implant Stability in Immediate Versus Early Implant Placement: A Randomized Controlled Clinical Trial
Brief Title: Assessment of Marginal Bone Loss and Anterior Implant Stability in Immediate Versus Early Implant Placement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yasser Ahmed (Other)
Responsible Party: Sponsor-Investigator, Yasser Ahmed, Associate Professor of Prosthodontics, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: IRB2023-H0113D-P-0494
Record Dates: First submitted 2025-05-15; First posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Marginal Bone Loss

STUDY DESIGN:
Intervention Model Description: split-mouth design
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate implant placement (Experimental)
  Interventions: Procedure: Immediate implant placement
- Early implant placement (Active Comparator)
  Interventions: Procedure: Early implant placement

INTERVENTIONS:
Procedure: Immediate implant placement — Tooth extraction was performed atraumatically on one side, followed by immediate implant placement, right after extraction.
  Arms: Immediate implant placement
Procedure: Early implant placement — The tooth was extracted, and the implant was placed four weeks later (early placement).
  Arms: Early implant placement

SUMMARY:
This study aims to determine the differences in implant stability and measurement of bone loss near implants between two different healing approaches used for teeth replacement in the front part of the upper jaw.

ELIGIBILITY:
Inclusion Criteria:

* Presence of unrestorable bilateral anterior teeth.
* Harmonious gingival contour and thick gingival phenotype
* Minimum 4 mm of apical bone and 2 mm of intact labial plate
* Absence of periapical pathology

Exclusion Criteria:

* Systemic conditions affecting osseointegration or healing
* Active oral infections or periodontal disease
* Dehiscence or fenestration defects
* Poor oral hygiene or heavy smoking

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Marginal Bone Loss | up to 12 months
  Cone beam computed tomography (CBCT) scans were obtained at the time of final restoration and post-placement. Measurements were made (in mm) from the implant platform to the most coronal bone level using OnDemand3D software. Each scan was oriented to align the implant with the axial plane. Measurements were performed by a single calibrated examiner to a precision of 0.01 mm.
Implant stability | up to 12 months
  Implant Stability Quotient (ISQ) values were measured using Osstell. To ensure accuracy, the probe was positioned at a 90° angle and 3 mm above soft tissue level, as recommended in previous protocols. Osstell's patented technology uses the ISQ scale, with values ranging from 1 to 100, where higher values indicate greater stability

CONTACTS AND LOCATIONS:
Locations (1):
- Beirut Arab University, Beirut, Lebanon